CLINICAL TRIAL: NCT04993118
Title: Effects Of Integrated Neuromuscular Inhibition Technique On Upper Trapezius Trigger Points In Patients With Non-Specific Neck Pain
Brief Title: Integration of Neuromuscular Inhibition Technique On Trapezius Trigger Points.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00770 Ammara Malik
Record Dates: First submitted 2021-04-10; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Myofascial Trigger Point Pain
Keywords: Neck pain; Trapezius trigger points; INIT
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Official Title: Effects of Integrated Neuromuscular Inhibition technique on upper trapezius trigger points in patients with non-specific neck pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Neuromuscular inhibition technique (Experimental): Experimental group received Integrated neuromuscular inhibition technique. At first ischemic compression was given using a pincer grip over the active trigger point till the tissue barrier was felt .The process was repeated till the tension reduced for 90 seconds.Ischemic compression was followed by the application of strain counterstrain. M If pain was reproduced the pressure was maintained over the active trigger point as the position of ease was identiﬁed. Once the position of ease was identiﬁed, it was held for 90 seconds and repeated for three to ﬁve repetitions. Muscle energy technique was applied as last part of iINIT.Each isometric contraction was held for 7-10 seconds and was followed by further contralateral side bending, ﬂexion, and ipsilateral rotation to maintain the soft tissue stretch. Each stretch was held for 30 seconds and was repeated three to ﬁve times per treatment session
  Interventions: Other: Integrated Neuromuscular Inhibition technique
- Ischemic Compression,Hotpack,TENS (Active Comparator): Control group received conventional physical therapy. It included HOT Packs ( 20 minutes) , TENS (10 minutes) ,Ischemic compression .Using a pincer grasp, we identified the trigger point. Once the trigger point was identiﬁed we applied ischemic compression by placing the thumb and index ﬁnger over the active TrP. Slow, increasing levels of pressure was applied until the tissue resistance barrier was identiﬁed. Pressure was maintained until a release of the tissue barrier was felt. At that time, pressure was again applied until a new barrier was felt. This process was repeated until tension/tenderness is unable to be identiﬁed
  Interventions: Other: Ischemic Compression,Hotpack,TENS

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition technique — Integrated Neuromuscular inhibition technique At first ischemic compression was given using a pincer grip over the active trigger point till the tissue barrier was felt .The process was repeated till the tension reduced for 90 seconds.Ischemic compression was followed by the application of strain counterstrain. Once the position of ease was identiﬁed, it was held for 90 seconds and repeated for three to ﬁve repetitions. Muscle energy technique was applied as last part of integrated neuromuscular inhibition technique . Each isometric contraction was held for 7-10 seconds and was followed by further contralateral side bending, ﬂexion, and ipsilateral rotation to maintain the soft tissue stretch. Each stretch was held for 30 seconds and was repeated three to ﬁve times per treatment session
  Arms: Integrated Neuromuscular inhibition technique
Other: Ischemic Compression,Hotpack,TENS — Control group received conventional physical therapy. It included HOT Packs ( 20 minutes) , TENS (10 minutes) ,Ischemic compression .Using a pincer grasp, we identified the trigger point. Once the trigger point was identiﬁed we applied ischemic compression by placing the thumb and index ﬁnger over the active TrP. Slow, increasing levels of pressure was applied until the tissue resistance barrier was identiﬁed. Pressure was maintained until a release of the tissue barrier was felt. At that time, pressure was again applied until a new barrier was felt. This process was repeated until tension/tenderness is unable to be identiﬁed
  Arms: Ischemic Compression,Hotpack,TENS

SUMMARY:
The purpose of the study is to find the effects of integrated neuromuscular inhibition technique on upper trapezius trigger points in patients with non specific neck pain. A randomized control trial was conducted at Iqbal hospital. The sample size was 24calculated through open-epitool.But 30 patients were added in the study to increase the statistical power of analysis.The participants were divided into two interventional groups each having 15 participants. The study duration was six months. Sampling technique applied was Purposive sampling for recruitment and group randomization using sealed envelope method. Only 25 to 45 years participants (both male and female) with upper trapezius trigger points and non specific neck pain of less than 3 months were included in the study. Tools that were used in this study are NDI questionnaire, NPRS and inclinometer. Data was collected at baseline , 2nd and 4th of treatment. Data was analyzed through SPSS version 20.

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal disorder. The cause of neck pain is variable and can result from specific musculoskeletal conditions, infections, inflammatory conditions, trauma, rheumatic diseases, or congenital diseases. When neck pain is not attributed to a specific pathology, and is of a vague musculoskeletal origin which is difficult to identify, the condition is labelled non-specific. Up to 67% of world's population may present with non-specific neck pain at least once in their lives. Although the duration and course of the pain may vary, most patients experience chronic or recurrent pain. Evidence suggests that myofascial trigger points are commonly present in patients with non specific neck pain.

The myofascial trigger point ''a hyperirritable spot, usually within a taut band of skeletal muscle or in the muscle fascia which is painful on compression and can give rise to characteristic referred pain, motor dysfunction, and autonomic phenomena. Patients may have regional ,persistent pain resulting in decreased range of motion in the affected muscles. Trigger points may develop after an initial injury to muscle fibers. This injury may include a noticeable traumatic event or repetitive micro trauma to the muscles. The trigger point causes pain and stress in the muscle or muscle fiber. As the stress increases, the muscles become fatigued and more susceptible to activation of additional trigger points. When predisposing factors combine with a triggering stress event, activation of a trigger point occurs. This theory is known as the ''injury pool theory'.

Trigger points are classified as active or latent. Active myofascial trigger point is spontaneously painful and gives rise to a number of well described symptoms: local and/or referred pain; muscle weakness and tightness. Latent myofascial trigger points on the other hand, are generally considered minor, sub-clinical neuromuscular lesions that are pain-free unless compressed though shown to be associated with increased sensitivity to muscle stretch, decreased strength. In the upper quadrant, postural muscles, in general, and the upper trapezius , in particular, are most affected by trigger points .It extends from the external protuberance of the occipital bone to the lower thoracic vertebrae and laterally to the spine of the scapula. The trapezius has upper, middle, and lower groups of fibers. Neck pain is provoked by trigger points of trapezius.Patients with trigger points of trapezius usually present with neck pain,decreased cervical range of motion,tightness of trapezius Various treatment techniques that are utilized for treating trigger points are LASER , dry needling, ultrasound, TENS, trigger point pressure release /ischemic compression, muscle energy technique , myofascial release therapy , positional release therapy i.e. strain counter strain technique and integrated neuromuscular inhibitory technique.The integrated neuromuscular inhibition technique is a manual deactivation trigger points technique and includes the application of ischemic compression, muscle energy technique and strain counter strain technique. Ischemic compression ('inhibition') is applied to an active trigger point by means of direct finger or thumb pressure until local or referred pain begins to modify. Following this, the tissues in which the trigger point lies are positioned in such a way as to modify the pain . After 90 seconds the patient is asked to introduce an isometric contraction into the tissues and to hold this for 7-10 seconds. This recruits the precise fibers which had been repositioned to obtain the positional release. These previously hypertonic or fibrotic tissues are then stretched so that the specifically targeted fibers are lengthened. A rhythmic activation of antagonist muscles in a series of 'pulsed' contractions is a useful final stage of this sequence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non specific neck pain < 3 months duration
* Patients who have TrPs in upper trapezius confirmed on basis of Travel and Simons diagnostic criteria

Exclusion Criteria:

* • Patients having any trauma

  * Signs of any serious pathology ( e.g malignancy, inflammatory disorder or fracture)
  * Signs of spinal cord compression
  * Signs of nerve root involvement
  * History of neck surgery in previous 12 months
  * History of cervical degenerative joint disease
  * Autoimmune conditions

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 months
  Neck Disability Index (NDI) questionnaire ( for measuring neck disability). Total score 50,minimum score is 0 and maximu,m score is 50 parameter minimum and max
Numeric Pain Rating Scale | 6 months
  NPRS, for measuring pain intensity.minimum score is o and maximum is 10

SECONDARY OUTCOMES:
range of motion (Cervical flexion) | 6 months
  inclinometer(For measuring flexion range of motion)
range of motion (Cervical extention) | 6 months
  inclinometer(for measuring extension range of motion)
range of motion (Cervical side bending,right left ) | 6 months
  inclinometer(for measuring cervical side bending range of motion)
range of motion (Cervical rotation right left,) | 6 months
  inclinometer(for measuring cervical rotation range of motion)

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Iqbal Hospital, Attock, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagrale AV, Glynn P, Joshi A, Ramteke G. The efficacy of an integrated neuromuscular inhibition technique on upper trapezius trigger points in subjects with non-specific neck pain: a randomized controlled trial. J Man Manip Ther. 2010 Mar;18(1):37-43. doi: 10.1179/106698110X12595770849605. PMID 21655422
- [Background] Sarigiovannis P, Hollins B. Effectiveness of manual therapy in the treatment of non-specific neck pain: a review. Physical therapy reviews. 2005;10(1):35-50.
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del-Moral O, Pacheco-da-Costa S, Prieto-Merino D, Sanchez-Sanchez B. Health related quality of life improvement in chronic non-specific neck pain: secondary analysis from a single blinded, randomized clinical trial. Health Qual Life Outcomes. 2018 Nov 6;16(1):207. doi: 10.1186/s12955-018-1032-6. PMID 30400984
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Miangolarra JC. Myofascial trigger points in subjects presenting with mechanical neck pain: a blinded, controlled study. Man Ther. 2007 Feb;12(1):29-33. doi: 10.1016/j.math.2006.02.002. PMID 21882489
- [Background] Vincent K, Maigne JY, Fischhoff C, Lanlo O, Dagenais S. Systematic review of manual therapies for nonspecific neck pain. Joint Bone Spine. 2013 Oct;80(5):508-15. doi: 10.1016/j.jbspin.2012.10.006. Epub 2012 Nov 16. PMID 23165183
- [Background] Blikstad A, Gemmell H. Immediate effect of activator trigger point therapy and myofascial band therapy on non-specific neck pain in patients with upper trapezius trigger points compared to sham ultrasound: a randomised controlled trial. Clinical Chiropractic. 2008;11(1):23-9.
- [Background] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Background] Shah JP, Danoff JV, Desai MJ, Parikh S, Nakamura LY, Phillips TM, Gerber LH. Biochemicals associated with pain and inflammation are elevated in sites near to and remote from active myofascial trigger points. Arch Phys Med Rehabil. 2008 Jan;89(1):16-23. doi: 10.1016/j.apmr.2007.10.018. PMID 18164325
- [Background] Lucas KR, Rich PA, Polus BI. Muscle activation patterns in the scapular positioning muscles during loaded scapular plane elevation: the effects of Latent Myofascial Trigger Points. Clin Biomech (Bristol). 2010 Oct;25(8):765-70. doi: 10.1016/j.clinbiomech.2010.05.006. Epub 2010 Jul 27. PMID 20667633
- [Background] Hwang UJ, Kwon OY, Yi CH, Jeon HS, Weon JH, Ha SM. Predictors of upper trapezius pain with myofascial trigger points in food service workers: The STROBE study. Medicine (Baltimore). 2017 Jun;96(26):e7252. doi: 10.1097/MD.0000000000007252. PMID 28658117
- [Background] Sibby GM, Kavitha Vishal S. Effectiveness of integrated neuromuscular inhibitory technique and LASER with stretching in the treatment of upper trapezius trigger points. Journal of exercise science and physiotherapy. 2009;5(2):115.
- [Background] Gemmell H, Allen A. Relative immediate effect of ischaemic compression and activator trigger point therapy on active upper trapezius trigger points: A randomised trial. Clinical Chiropractic. 2008;11(4):175-81.
- [Background] Saadat Z, Hemmati L, Pirouzi S, Ataollahi M, Ali-Mohammadi F. Effects of Integrated Neuromuscular Inhibition Technique on pain threshold and pain intensity in patients with upper trapezius trigger points. J Bodyw Mov Ther. 2018 Oct;22(4):937-940. doi: 10.1016/j.jbmt.2018.01.002. Epub 2018 Jan 17. PMID 30368338
- [Background] Mehdikhani R, Okhovatian F. RETRACTED: Immediate effect of muscle energy technique on latent trigger point of upper trapezius muscle. Elsevier; 2012.
- [Background] Sharma A, Angusamy R, Kalra S, Singh S. Efficacy of post-isometric relaxation versus integrated neuromuscular ischaemic technique in the treatment of upper trapezius trigger points. Indian Journal of Physiotherapy and Occupational Therapy. 2010;4(3):1-5.
- [Background] NEELIMA A. TO ASSESS THE EFFECTIVENESS OF INTEGRATED NEURO MUSCULAR INHIBITORY TECHNIQUES (INIT) WITH STABILIZATION EXERCISES VERSUS ULTRASOUND WITH STABILIZATION EXERCISES ON UPPER TRAPEZIUS TRIGGERPOINTS IN MYOFASCIAL PAIN SYNDROME 2013.
- [Background] Mobilization INI. Comparison of the effect of spinal accessory nerve mobilization, integrated neuromuscular inhibition technique and conventional therapy on in upper trapezius trigger point. Quadriceps Femoris Strength Training: effect of Neuromuscular Electrical Stimulation Vs Isometric Exercise in Osteoarthritis of Knee. 2015;9(3):135.
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Bush KW, Collins N, Portman L, Tillett N. Validity and intertester reliability of cervical range of motion using inclinometer measurements. Journal of Manual & Manipulative Therapy. 2000;8(2):52-61.
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888
- [Background] Aggarwal S, Bansal G. Efficacy of integrated neuromuscular inhibition technique in improving cervical function by reducing the trigger points on upper trapezius muscle: A randomized controlled trial. Muller Journal of Medical Sciences and Research. 2018;9(1):1-.
- [Background] Farina S, Casarotto M, Benelle M, Tinazzi M, Fiaschi A, Goldoni M, Smania N. A randomized controlled study on the effect of two different treatments (FREMS AND TENS) in myofascial pain syndrome. Eura Medicophys. 2004 Dec;40(4):293-301. PMID 16175154